CLINICAL TRIAL: NCT01385488
Title: Bioelectrical Impedance for Self-monitoring of Breast Cancer Related Lymphedema
Brief Title: Bioelectrical Impedance for Self-monitoring of Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Sheila Ridner, professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 110032
Record Dates: First submitted 2011-04-28; First posted 2011-06-30 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Lymphedema
Keywords: lymphedema; breast cancer; self care; bioelectrical impedance; monitoring
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-monitoring (Experimental): participants will use bioelectrical impedance to self-monitor arm volume at home
  Interventions: Behavioral: self-monitor arm volume
- completion of forms (No Intervention): participants will complete self-report forms

INTERVENTIONS:
Behavioral: self-monitor arm volume — bioelectrical impedance
  Arms: self-monitoring

SUMMARY:
* Breast cancer treatment-related lymphedema requires life-long self-care is required.
* No objective measurement mechanism exists that can easily be used to self-monitor arm volume.
* Bioelectrical impedance devices approved for lymphedema measurement may be able to be used for self-monitoring.
* The investigators will conduct a two-part study to first develop an impedance driven self-measurement protocal and then test the protocol in home settings.
* The investigators hypothesize in part two of the study that when compared to participants who are not self-monitoring, those who self-monitor limb volume will: 1) report more days of garment use, skin care, and simple-MLD; and, 2) have fewer, less distressful, less intense symptoms, better productivity/activity, report higher perceived self-management/self-efficacy and QOL; experience fewer missed days of work, lymphedema treatment days, arm infections, and have a smaller number of antibiotic prescriptions.

DETAILED DESCRIPTION:
Breast cancer treatment-related lymphedema (swelling) is an incurable, chronic condition experienced by a significant percentage of breast cancer survivors. It has many associated symptoms, negatively impacts quality of life (QOL), and increases health care costs. As with other chronic diseases, such as diabetes, life-long self-care is required. No objective measurement mechanism exists that can easily be used to self-monitor arm volume, a key self-care outcome. Those with lymphedema are forced to rely on visual recognition of increasing volume to know if their self-care is effective and when to seek treatment. Timely recognition of worsening swelling is believed to result in better patient outcomes; however, substantial volume increases often occur before observable changes are noted and this window of opportunity is missed. Many with lymphedema only seek care when they have developed infection in the swollen limb.

The inability to objectively monitor arm volume on a regular basis likely results in discomfort, poorer QOL, and increased health care costs.The broad, long-term objective of this application is to develop a method for monitoring arm lymphedema that can be used at home to improve lymphedema self-management and patient outcomes. To accomplish this, the investigators will conduct a two-phase, translational pilot study to explore the use of a hand-held bioelectrical impedance device as an arm volume self-measurement method.

The purpose of Phase 1 is to develop a bioelectrical impedance self-measurement protocol. Healthy volunteers (n=11) and individuals with lymphedema (n=11) will be in Phase 1 (protocol development). This will take place in laboratory and home settings. This Phase is not interventional and is not detailed in this posting.

The purpose of Phase 2 is to compare self-care activities and health and economic outcomes between breast cancer survivors with lymphedema following the self-monitoring protocol developed in Phase 1 and breast cancer survivors with lymphedema not on protocol (n=42).The protocol will be field-tested by breast cancer survivors with lymphedema in Phase 2 (a two group randomized clinical trial). One group will self-measure with impedance at home for three months, weekly record self-care activities, and will complete follow-up assessments. The other group will mirror Group 1 except for impedance measurements. This is an interventional study and is presented as such in this clinical trial posting.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Volunteers for Phase 1: no known history of cancer or lymphatic disease.
2. Lymphedema volunteers Phases 1 &2: history of breast cancer and diagnosis of lymphedema in one arm.
3. All volunteers: ≥ 21 years of age.

Exclusion Criteria:

1. Healthy Volunteers Phase 1: history of arm surgery or family history of primary lymphedema.
2. Lymphedema volunteers Phases 1 & 2: bilateral lymphedema.
3. All volunteers:

   * inability to stand upright;
   * conditions that could cause swelling: pregnancy, congestive heart failure, liver failure;
   * infection, open sores on arms, or known sensitivity to electrodes;
   * pacemakers or internal defibrillators;
   * currently undergoing IV chemotherapy or radiation; or
   * use of laxatives or diuretics to lose weight.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
self care behaviors | 4 months
  individual tasks initiated by a participant to care for their lymphedema that may vary from participant to participant.
Self-care self efficacy | 4 months
  perception of abilty to provide lymphedema self-care

SECONDARY OUTCOMES:
health | four months
  lymphedema associated symptoms
quality of life | 4 months
  quality of life
economics | 4 months
  expense in terms of lost income or out-of pocket payments related to lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila H Ridner, PHD, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Vanderbilt Univeristy School Of Nursing, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided